CLINICAL TRIAL: NCT04749069
Title: The Comparison of Two Different Techniques of Remifentanil Consumption During Implantable Vascular Access Device Procedures
Brief Title: Anesthesia for Vascular Access Devices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kartal Kosuyolu Yuksek Ihtisas Education and Research Hospital (Other Government)
Collaborators: Trakya University (Other)
Responsible Party: Principal Investigator, Ayse Baysal, The comparison of patient-controlled sedation method and anesthesiologist-controlled sedation method in port interventions, Kartal Kosuyolu Yuksek Ihtisas Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2012.3.35(#)
Record Dates: First submitted 2021-02-04; First posted 2021-02-10 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Opioid Use, Unspecified; Remifentanil; Sedation Complication; Analgesia; Satisfaction, Patient; Vascular Access Complication
MeSH Terms: conditions — Agnosia; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: This is a prospective, single-blinded randomized clinical study. The patients were divided into two groups with the method of one to one allocation and with the use of sealed envelope randomization.The first group was continuous infusion group (Group CI) and intravenous continuous remifentanil was infused after starting at a dosage of 0.1 µg/kg/min and the dose was raised incrementally up to 1µg/kg/min if required. The second group was intravenous bolus patient-controlled sedation analgesia (PCSA) and remifentanil infusion at a dose of 0.05 µg/kg, bolus of 0.1 μg/kg with lock-out time of three minutes was used. In both groups, a bolus dose of 0.1 µg/kg remifentanil was administered. The data evaluated include; level of pain and sedation, total amount of remifentanil consumption, bolus doses of remifentanil, use of a rescue medication, patient and surgeon satisfaction, hemodynamic data and adverse events.
Who Masked: Participant, Outcomes Assessor
Masking Description: In our study, random allocation sequence was performed using a computer programme for each patient to prevent bias. For concealed allocation, patients were randomly allocated into one group using a numbered, opaque and sealed envelope. A randomized block design is as follows: code A was given to the first group, and code B was given to the second group. The participant, data collector and data analyzer were blinded. This study was a single-blinded controlled study because the sedation and analgesia were administered by anesthesiology residents who were unaware of the technique and the study protocol however, the protocol was known by the experienced anesthesiologist who was attending the case and collecting the data during the procedure. The preparation of remifentanil solutions and installation of the infusion devices were done by an anesthesiologist who was blinded for the study groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Continuous infusion of remifentanil (Experimental): In continuous infusion group of patients, remifentanil was infused at a dose of 0.1 µg/kg/min and the additional bolus dose of 0.1 µg/kg was given if required. Before start of the operation, in both groups of patients, intravenous remifentanil at a bolus dose of 0.1 µg/kg was administered slowly in a duration of 60 seconds.
  Interventions: Diagnostic Test: Comparison of pain intensity rating scale
- Patient-controlled sedoanalgesia (PCSA) of remifentanil (Experimental): In PCSA group of patients, remifentanil was given by bolus PCSA using a pump (Pain Management Provider, Abbott Laboratories and Eczacibasi-Baxter, Ireland). In PCSA group of patients, remifentanil infusion was at a dose of 0.05 µg/kg, a bolus dose of 0.1 μg/kg with a lock-out time of three minutes.
  Interventions: Diagnostic Test: Comparison of pain intensity rating scale

INTERVENTIONS:
Diagnostic Test: Comparison of pain intensity rating scale — Comparison of numerical pain intensity rating scale Comparison of faces pain rating scale Comparison of consumption of total amount of remifentanil
  Other Names: Sedation-Numerical pain intensity rating scale, Faces pain rating scale; Analgesia-Ramsey sedation scale; Drug-Remifentanil consumption of total amount of remifentanil

SUMMARY:
Our aim was to investigate whether remifentanil use in both infusion and bolus techniques could provide sufficient sedation and analgesia without serious adverse effects for central venous access device procedures under monitored anesthesia care.

DETAILED DESCRIPTION:
The insertion and removal of implantable venous access devices (port-a-cath type) requires moderate level of sedation and monitored anesthesia care to prevent pain and anxiety of patients during the procedure. According to the American Society of Anesthesiologist Physical Status Score, monitored anesthesia care is a planned procedure where a patient undergoes local anesthetic infiltration together with sedation and analgesia. Remifentanil is a potent synthetic opioid with novel pharmacokinetic properties, including very rapid onset and an ultra short duration of action, making it effective for pain relief in short procedures. Remifentanil can be administered as either one of the techniques of intravenous continuous infusion (CI) or intravenous bolus patient-controlled sedation analgesia (PCSA).In previous studies, the insertion or removal of venous access procedures required either local anesthesia or low doses of orally administered anxiolytic medication. The infusion of remifentanil may cause respiratory depression and analgesic efficacy and safety of administration of remifentanil infusion and/or bolus doses of remifentanil during the administration of one of the techniques of either CI or PCSA in short term procedures has not been well studied. The prospective trials that compare analgesic efficacy and adverse events related to intravenous remifentanil consumption in sedation and analgesia of short procedures are very limited.

This study aims to compare level of pain and sedation, total amount of remifentanil consumption, bolus doses of remifentanil, patient and surgeon satisfaction, hemodynamic data and adverse events of two different techniques of intravenous remifentanil use such as; intravenous continuous infusion (CI) or intravenous bolus patient-controlled sedation analgesia (PCSA) in patients under moderate level of sedation for vascular access procedures.

ELIGIBILITY:
Inclusion Criteria:

1. 30-80 years old,
2. American Society of Anesthesiologists Physical Status I to III,
3. Referred for an venous access device implantation or removal procedure.

Exclusion Criteria:

1. morbid obesity (body mass index > 40),
2. severe asthma, chronic obstructive lung disease, diabetes mellitus, hepatorenal disease,
3. a history of opioid allergy,
4. long-term opioid use or chronic pain,
5. ASA PS ≥ 4,
6. presence of epilepsy,
7. acute cerebrovascular event,
8. presence of hemodynamical instability such as peripheral oxygen saturation < 90%, systolic blood pressure < 60 mmHg and heart rate ≤ 40 bpm,
9. patients complaining about intense pain before the procedure.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2012-08-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
The Numeric Pain Intensity Rating Scale (NPRS) | After incision and during operative time every five minutes, through the operative time period up to two hours of time.
  During NPRS pain evaluation, a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain comparison and this includes 0 as no pain and 10 as the worst pain imaginable. There is a comparison of pain scale scores as a decrease of pain relief in an amount of 30% from the pain at start between the two groups.
The faces pain rating scale | After incision and during operative time every five minutes, through the operative time period up to two hours of time.
  The scale shows a series of faces ranging from a happy face at 0, or "no hurt", to a crying face at 10, which represents "hurts like the worst pain imaginable".
Measurement of sedation and analgesia | After incision and during operative time every five minutes, through the operative time period up to two hours of time.
  The comparison of the use of Ramsay Sedation Scale for measurement of sedation and analgesia between the two groups.The Ramsay Sedation Scale involves 6 levels and these include; 1- Patient is anxious and agitated or restless, or both, 2- Patient is co-operative, oriented, and tranquil, 3-Patient responds to commands only, 4- Patient exhibits brisk response to light glabellar tap or loud auditory stimulus, 5-Patient exhibits a sluggish response to light glabellar tap or loud auditory stimulus, 6- Patient exhibits no response.

SECONDARY OUTCOMES:
Total Remifentanil Consumption | At the end of operation, through the operative time period up to two hours of time.
  The comparison of the use of total remifentanil consumption between the two groups.
Modified Aldrete Score | Through the recovery room time period before discharge up to one hour time.
  The comparison of the use of Modified Aldrete scores in the recovery room before discharge between the two groups.
Duration of operation | At the end of operation, through the operative time period up to two hours of time.
  The comparison of the duration of operations between the two groups.
Incidence of adverse events and side effects. | After operation in the recovery room through the recovery room time period before discharge up to one hour time and 24 hour after surgery.
  The comparison of the incidence of adverse events and side effects between the two groups.
Patient and surgeon satisfaction | The collection of questionnaire at the end of operation in recovery room after recovery from sedation in a total of ten minutes time.
  The comparison of satisfaction of patient and surgeon by a questionnaire at the end of operation between two groups.
Recovery time | Through the recovery room time period before discharge up to one hour time.
  The comparison of recovery time between two groups.
Systolic blood pressure values during operation and in the recovery room. | The collection of systolic blood pressure in mmHg unit values every 15 minutes through the operative time period up to two hours of time and through the recovery room time period before discharge up to one hour time
  The comparison of systolic blood pressure values during operation and in the recovery room between two groups.
Diastolic blood pressure values during operation and in the recovery room. | The collection of diastolic blood pressure in mmHg unit values every 15 minutes through the operative time period up to two hours of time and through the recovery room time period before discharge up to one hour time
  The comparison of diastolic blood pressure values during operation and in the recovery room between two groups.
Heart rate values during operation and in the recovery room. | Through the operative time period up to two hours of time and through the recovery room time period before discharge up to one hour time.
  The comparison of heart rate values during operation and in the recovery room between two groups.
Pulse oximetry values during operation and in the recovery room. | hrough the operative time period up to two hours of time and through the recovery room time period before discharge up to one hour time
  The comparison of Pulse oximetry values during operation and in the recovery room between two groups.
Hospital Stay | Through the duration of stay in hospital before discharge up to seventy two hours time.
  The comparison of hospital stay between two groups.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Trakya University Faculty of Medicine Department of Anesthesiology, Edirne
  - Kartal Kosuyolu High Speciality Training and Research Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: Yes
Purpose: The aim was to compare analgesic efficacy and adverse effects of two different techniques of intravenous remifentanil consumption in patients undergoing vascular access device procedures with monitored anesthesia care. The data evaluated include; level of pain and sedation, total amount of remifentanil consumption, bolus doses of remifentanil, patient and surgeon satisfaction, hemodynamic data and adverse events.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The data will become available after registration and will be available upon request from the Clinical Study Director at any time after registration.
Access Criteria: Study Protocol and Statistical Package for the Social Sciences computer program data.

REFERENCES:
- [Background] Honarmand A, Safavi M, Nemati K, Oghab P. The efficacy of different doses of Midazolam added to Lidocaine for upper extremity Bier block on the sensory and motor block characteristics and postoperative pain. J Res Pharm Pract. 2015 Jul-Sep;4(3):160-6. doi: 10.4103/2279-042X.162359. PMID 26312256
- [Background] Hinkelbein J, Lamperti M, Akeson J, Santos J, Costa J, De Robertis E, Longrois D, Novak-Jankovic V, Petrini F, Struys MMRF, Veyckemans F, Fuchs-Buder T, Fitzgerald R. European Society of Anaesthesiology and European Board of Anaesthesiology guidelines for procedural sedation and analgesia in adults. Eur J Anaesthesiol. 2018 Jan;35(1):6-24. doi: 10.1097/EJA.0000000000000683. PMID 28877145
- [Background] Ryu JH, So YM, Hwang JW, Do SH. Optimal target concentration of remifentanil during cataract surgery with monitored anesthesia care. J Clin Anesth. 2010 Nov;22(7):533-7. doi: 10.1016/j.jclinane.2010.02.007. PMID 21056810
- [Result] Sun GQ, Gao BF, Li GJ, Lei YL, Li J. Application of remifentanil for conscious sedation and analgesia in short-term ERCP and EST surgery. Medicine (Baltimore). 2017 Apr;96(16):e6567. doi: 10.1097/MD.0000000000006567. PMID 28422846
- [Result] Chang DH, Hiss S, Herich L, Becker I, Mammadov K, Franke M, Mpotsaris A, Kleinert R, Persigehl T, Maintz D, Bangard C. Implantation of venous access devices under local anesthesia: patients' satisfaction with oral lorazepam. Patient Prefer Adherence. 2015 Jul 7;9:943-9. doi: 10.2147/PPA.S80330. eCollection 2015. PMID 26185424
- [Result] Zanvettor A, Lederer W, Glodny B, Chemelli AP, Wiedermann FJ. Procedural sedation and analgesia for percutaneous trans-hepatic biliary drainage: Randomized clinical trial for comparison of two different concepts. Open Med (Wars). 2020 Aug 28;15(1):815-821. doi: 10.1515/med-2020-0220. eCollection 2020. PMID 33336039
- [Result] Fanti L, Agostoni M, Gemma M, Gambino G, Facciorusso A, Guslandi M, Torri G, Testoni PA. Remifentanil vs. meperidine for patient-controlled analgesia during colonoscopy: a randomized double-blind trial. Am J Gastroenterol. 2009 May;104(5):1119-24. doi: 10.1038/ajg.2009.53. Epub 2009 Mar 31. PMID 19337241
- [Result] Vardon Bounes F, Pichon X, Ducos G, Ruiz J, Samier C, Silva S, Sommet A, Fourcade O, Conil JM, Minville V. Remifentanil for Procedural Sedation and Analgesia in Central Venous Catheter Insertion: A Randomized, Controlled Trial. Clin J Pain. 2019 Aug;35(8):691-695. doi: 10.1097/AJP.0000000000000725. PMID 31094935